CLINICAL TRIAL: NCT07261930
Title: Effectiveness of Preoperative Intravenous Tranexemic Acid on Reduction of Perioperative Blood Loss in Open Intramedullary Nail Fixation of Femoral Shaft Fractures in Mulago
Brief Title: Effectiveness of Tranexamic Acid in Reducing Blood Loss During Femoral Nail Surgery
Acronym: TXA-FemNail
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Masaka Regional Referral Hospital (Other Government)
Collaborators: Mulago Hospital, Uganda (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Kabazzi Kaweesa Paul, Principle Investigator, Masaka Regional Referral Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MskRRH-ORTHO-2025-001
Record Dates: First submitted 2025-07-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Femoral Fractures; Hemorrhage, Surgical; Tranexamic Acid Use
Keywords: Femoral Shaft Fractures; Intramedullary Nailing; Perioperative Hemorrhage; Tranexamic Acid; Orthopedic Surgery; Blood Loss, Surgical; Blood Transfusion; Open Reduction and Internal Fixation; Developing Countries
MeSH Terms: conditions — Femoral Fractures; Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label prospective cohort study where all enrolled participants receive the same intervention - a preoperative intravenous dose of tranexamic acid (15 mg/kg) prior to open intramedullary nailing of femoral shaft fractures. There is no control or comparison group within the trial; outcomes are assessed against pre-defined benchmarks or historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm: IV TXA Before Femoral Nailing (Experimental): Participants in this arm received a single preoperative intravenous dose of tranexamic acid (Kapron®, Amoun Pharma, Egypt) at 15 mg/kg, administered slowly over 10 minutes approximately 10 minutes before skin incision. The intervention was intended to reduce perioperative blood loss in patients undergoing open intramedullary nail fixation of isolated femoral shaft fractures at Mulago National Referral Hospital, Uganda. All participants received standard perioperative care, including preoperative antibiotics and anesthesia. No control or placebo group was included in this single-arm, open-label study.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous tranexamic acid (Kapron®, Amoun, Egypt) administered as a single dose of 15 mg/kg, diluted in normal saline and given slowly over 10 minutes, approximately 10 minutes prior to skin incision. The drug was supplied in 500 mg/5 mL ampoules and administered by the anesthetist in the operating theater. This intervention was given once before surgery in patients undergoing open intramedullary nail fixation of isolated femoral shaft fractures. No additional doses or postoperative administration of TXA were used.
  Other Names: Kapron

SUMMARY:
This clinical study aims to evaluate the safety and effectiveness of administering a single intravenous dose of tranexamic acid (TXA) before surgery to reduce blood loss in patients undergoing open intramedullary nailing for femoral shaft fractures. In many resource-limited settings, including Uganda, this surgical approach is common due to lack of fluoroscopic equipment, and it is known to be associated with significant perioperative blood loss.

Tranexamic acid is an antifibrinolytic agent that helps stabilize blood clots and is widely used to reduce bleeding in major surgeries such as joint replacements and spinal procedures. However, its role in trauma-related open femoral surgeries in low-resource settings remains underexplored.

This study investigates whether preoperative intravenous TXA can safely reduce blood loss and transfusion needs during and after surgery in patients with isolated femoral shaft fractures managed at Mulago National Referral Hospital.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm cohort study designed to assess the safety and effectiveness of preoperative intravenous tranexamic acid (TXA) in adult patients undergoing open intramedullary nailing for femoral shaft fractures in a resource-limited hospital setting.

The study enrolled 43 adult participants with isolated, closed femoral shaft fractures scheduled for surgical fixation at Mulago National Referral Hospital. Each participant received a single dose of intravenous tranexamic acid (15 mg/kg), administered over 10 minutes approximately 10 minutes prior to skin incision. The dose was prepared and delivered by the anesthetist in the operating theatre.

The primary objective of the study is to estimate perioperative blood loss, assessed by comparing preoperative hemoglobin concentration (taken 2 hours before surgery) to postoperative hemoglobin (taken 72 hours after surgery). Secondary objectives include assessing the proportion of patients requiring blood transfusions and documenting any adverse events associated with TXA administration, such as hypotension, nausea, or allergic reactions.

Surgical procedures were performed using either antegrade or retrograde open intramedullary nailing techniques. Standard perioperative care was provided, including preoperative antibiotics and either spinal or general anesthesia. All blood draws were conducted under aseptic conditions. Transfusion decisions followed standard clinical protocols based on clinical signs and hemoglobin thresholds.

This study is intended to inform clinical practice in low-resource settings by providing data on the potential utility of tranexamic acid in orthopedic trauma surgery where blood conservation is especially critical.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Patients with isolated, closed femoral shaft fractures
* Scheduled for open intramedullary nail fixation at Mulago National Referral Hospital
* Able and willing to provide written informed consent

Exclusion Criteria:

* Injury duration of more than one month
* Patients undergoing repeat surgery for a femoral fracture
* Pathological fractures of the femur
* Patients undergoing ORIF for more than one fracture during the perioperative period
* Known allergy to tranexamic acid
* History of bleeding disorders
* Presence of significant medical comorbidities (e.g., diabetes mellitus, history of deep vein thrombosis, or pulmonary embolism)
* Current use of anticoagulant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin Concentration from Preoperative to 72 Hours Postoperative | From 2 hours before surgery to 72 hours after surgery
  Hemoglobin concentration (g/dL) was measured 2 hours before surgery and again 72 hours after surgery. The difference between these two values was used to estimate total perioperative blood loss.

SECONDARY OUTCOMES:
Proportion of Patients Requiring Perioperative Blood Transfusion | From 2 hours before surgery to 72 hours after surgery
  The percentage of patients who received a blood transfusion during the perioperative period following administration of preoperative intravenous tranexamic acid (15 mg/kg). Blood transfusion indications were based on standardized clinical criteria and hemoglobin thresholds.
Incidence and Profile of Adverse Events Following Tranexamic Acid Administration | From 2 hours before surgery to 72 hours after surgery
  Capture and categorize any adverse events or side effects observed following the administration of intravenous tranexamic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kabazzi, Principal Investigator — Masaka Regional Referral Hospital
Locations (1):
- Mulago National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD) from this study due to limitations in data anonymization resources, ethical considerations, and the absence of prior consent for data sharing from participants. Additionally, the study was conducted in a single-center setting without provisions for long-term data storage or public data access infrastructure. Future data sharing may be considered upon request and subject to ethical review and approval.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT07261930/Prot_SAP_ICF_000.pdf